CLINICAL TRIAL: NCT01019434
Title: Radiation Therapy and Concurrent Plus Adjuvant Temsirolimus (CCI-779) Versus Chemo-Irradiation With Temozolomide in Newly Diagnosed Glioblastoma Without Methylation of the MGMT Gene Promoter - A Randomized Multicenter, Open-Label, Phase II Study.
Brief Title: Radiation Therapy and Temsirolimus or Temozolomide in Treating Patients With Newly Diagnosed Glioblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-26082-22081; EORTC-26082; EORTC-22081; EU-20987; 2008-003003-31 (EudraCT Number)
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma | interventions — Temozolomide; temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Temozolomide (Other): TMZ will be given at 75 mg/m2 daily for the whole period of RT including weekends as registered.
  Interventions: Drug: temozolomide
- Temsirolimus (Experimental): CCI-779 will be given i.v. once every week at 25 mg. Each treatment should be preceded by supportive medication with a histamine H2-receptor antagonist. A first dose of CCI-779, being 25 mg, will be given on day -7 from RT start.
  Interventions: Drug: temsirolimus

INTERVENTIONS:
Drug: temozolomide — TMZ will be given at 75 mg/m2 daily for the whole period of RT including weekends as registered.
  Arms: Temozolomide
Drug: temsirolimus — CCI-779 will be given i.v. once every week at 25 mg. Each treatment should be preceded by supportive medication with a histamine H2-receptor antagonist. A first dose of CCI-779, being 25 mg, will be given on day -7 from RT start.
  Arms: Temsirolimus

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Temsirolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. It is not yet known whether radiation therapy is more effective when given together with temsirolimus or temozolomide in treating patients with glioblastoma.

PURPOSE: This randomized phase II trial is studying giving radiation therapy together with temsirolimus to see how well it works compared with giving radiation therapy together with temozolomide in treating patients with newly diagnosed glioblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Document the activity profile of temsirolimus by the evaluation of overall survival at 1 year in patients with newly diagnosed glioblastoma multiforme, without methylation of the MGMT gene promoter, treated with temsirolimus before and concomitantly with radiotherapy, followed by temsirolimus maintenance therapy.

Secondary

* Investigate safety and tolerability of this therapy regimen in these patients.
* Assess progression-free survival and overall survival of these patients.
* Assess biomarkers in the tumor tissue relevant to temsirolimus and disease state, and their correlation to clinical outcome in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to institution, age in years (< 50 vs ≥ 50), Karnofsky performance status (PS) (< 80% vs ≥ 80%) OR ECOG PS (0 or 1 vs 2), and corticosteroid use (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Within 7 weeks after surgery or open biopsy, patients undergo radiotherapy 5 days a week for 6 weeks and receive oral temozolomide concurrently once daily for 6 weeks. Beginning 4 weeks after completion of concurrent chemoradiotherapy, patients receive adjuvant oral temozolomide once daily on days 1-5. Treatment with adjuvant temozolomide repeats every 28 days for up to 12 courses in the absence of disease progression and unacceptable toxicity.
* Arm II: Within 7 weeks after surgery or open biopsy, patients undergo radiotherapy 5 days a week for 6 weeks. Patients also receive temsirolimus IV over 30-60 minutes once weekly beginning 7 days before initiation of radiotherapy. After completion of chemoradiotherapy, patients receive maintenance temsirolimus IV once weekly in the absence of disease progression and unacceptable toxicity.

Frozen tumor biopsies or paraffin-embedded tumor material obtained from surgery or open biopsy and blood samples are collected for analysis of molecular markers, determination of the methylation status of the MGMT gene promoter (before randomization and at a later time), and other studies.

After completion of study therapy, patients are followed every 3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed (by open brain biopsy or from a neurosurgical resection of the tumor) supratentorial glioblastoma multiforme (GBM)

  * WHO grade IV disease
  * Newly diagnosed disease
* Must provide demonstration of an unmethylated MGMT-promoter
* At least 2 weeks and no more than 6 weeks since surgery or open biopsy
* Tumor tissue specimens (paraffin-embedded and/or frozen) from the GBM surgery or open biopsy must be available for central pathology review, MGMT status determination, and exploratory analysis of PI3-K/Akt/mTOR targets (P70S6K)

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 12 weeks
* WBC ≥ 3.0 x 10^9/L
* Absolute neutrophil count ≥ 1.5 x10^9/L
* Platelet count ≥ 75.0 x 10^9/L
* Hemoglobin ≥ 10.0 g/dL
* Bilirubin ≤ 1.5 times the upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2.5 x ULN
* AST and/or ALT ≤ 2.5 x ULN
* Serum creatinine < 1.5 x ULN
* PT and PTT normal
* Negative pregnancy test
* Not pregnant or nursing
* Fertile patients must use highly effective contraception
* No ischemic heart disease in the past 6 months
* 12-lead ECG normal
* No history of stroke
* No psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* No other malignancy within the past 5 years except adequately treated carcinoma in situ of the cervix or nonmelanoma skin cancer (with no subsequent evidence of recurrence)
* No serious concurrent systemic disorder including any of the following that, in the opinion of the investigator, would compromise the patient's ability to adhere to the protocol:

  * Active infection
  * HIV infection
  * Cardiac disease
  * QTc prolongation > 450/470 msec (males/females)
  * No patients with a congenital long-QT-syndrome in their own or family medical history, unless eligible at the investigator's discretion
* No known hypersensitivity to the study treatment
* No known hypersensitivity to antihistamines or other medical reason that prohibits the intake of antihistamines
* No current alcohol dependence or drug abuse
* No legal incapacity or limited legal capacity
* Able to undergo a gadolinium-enhanced MRI of the brain

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 4 weeks since prior and no concurrent investigational agent
* No prior stereotactic biopsy
* At least 30 days since prior drug therapy that has not received regulatory approval for any indication
* No chemotherapy within the past 5 years
* No prior chemotherapy for a brain tumor
* No prior radiotherapy to the head
* No other concurrent anticancer therapy
* No concurrent anticoagulation therapy except low-dose prophylactic low molecular weight heparin
* Concurrent steroid therapy allowed provided patient is on a stable or decreasing dose for ≥ 1 week
* At least 14 days since prior and no concurrent enzyme-inducing anticonvulsants (e.g., carbamazepine, phenobarbital, and phenytoin)
* No concurrent strong inducers or inhibitors of CYP3A4
* No concurrent planned surgery for other diseases (e.g., dental extraction)
* No placement of Gliadel® wafer during prior surgery

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2009-10; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Overall survival at 1 year | 1 year

SECONDARY OUTCOMES:
Percentages of worst Adverse Events or Laboratory Event grades as measured by CTCAEs Version 4.0 criteria | end of trial
Progression-free survival (PFS) probability at 6 months and at 12 months, and overall survival (OS) probability at 2 years | end of trial
Correlation between biomarkers relevant to temsirolimus and PFS and OS | end of trial

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Wick, Study Chair — Universitatsklinikum Heidelberg; Gianfranco Pesce, MD, Study Chair — Istituto Oncologico della Svizzera Italiana - Ospedale San Giovanni
Locations (13):
- UZ Leuven, Leuven, Belgium
- France (2):
  - Institut de Cancerologie de l'Ouest (ICO) - Centre Rene Gauducheau, Nantes-Saint Herblain
  - CHU Pitie-Salpetriere AP-HP, Paris
- Germany (2):
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Universitatsklinikum Heidelberg, Heidelberg
- Ospedale Bellaria, Bologna, Italy
- Netherlands (2):
  - Erasmus MC - Daniel den Hoed Cancer Center, Rotterdam
  - Medisch Centrum Haaglanden - Westeinde, The Hague
- ICO Badalona - Hospital Germans Trias i Pujol, Badalona, Spain
- Switzerland (2):
  - Ospedale Regionale Bellinzona e Valli, Bellinzona
  - UniversitaetsSpital Zuerich, Zurich
- United Kingdom (2):
  - Clatterbridge Cancer Centre NHS Foundation Trust, Bebington, Wirral
  - Western General Hospital, Edinburgh